CLINICAL TRIAL: NCT05124899
Title: Clinical Evaluation of the 80-Minute Water Resistant Sun Protection Factor (SPF) of Sunscreen Products According to the FDA Final Rule: Sunscreen Drug Products (2011)
Brief Title: Clinical Study to Evaluate the 80-Minute Water Resistant Sun Protection Factor (SPF) of Sunscreen Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 218007
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Results first posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2023-11

CONDITIONS: Sunscreening Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Only the outcomes (erythema) assessor is blinded to treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CAP UnScented (Experimental): Single topical application: 80 +/- 2 milligrams (mg) (2.0 +/- 0.05 mg per square centimeter [mg/cm^2]) of CAP UnScented will be applied to the assigned test site using a fingercot. Test material will be evenly spread over the test site using light pressure for 35 +/- 15 seconds.
  Interventions: Drug: CAP UnScented
- CAP Herbal Mint (Experimental): Single topical application: 80 +/- 2 mg (2.0 +/- 0.05 mg/cm^2) of CAP Herbal Mint will be applied to the assigned test site using a fingercot. Test material will be evenly spread over the test site using light pressure for 35 +/- 15 seconds.
  Interventions: Drug: CAP Herbal Mint
- CAP Mountain Berry (Experimental): Single topical application: 80 +/- 2 mg (2.0 +/- 0.05 mg/cm^2) of CAP Mountain Berry will be applied to the assigned test site using a fingercot. Test material will be evenly spread over the test site using light pressure for 35 +/- 15 seconds.
  Interventions: Drug: CAP Mountain Berry
- SPF Standard (Active Comparator): Single topical application: 80 +/- 2 mg (2.0 +/- 0.05 mg/cm^2) of SPF Standard will be applied to the assigned test site using a fingercot. Test material will be evenly spread over the test site using light pressure for 35 +/- 15 seconds.
  Interventions: Drug: SPF Standard Sunscreen

INTERVENTIONS:
Drug: CAP UnScented — Sunscreen lip balm.
  Arms: CAP UnScented
Drug: CAP Herbal Mint — Sunscreen lip balm.
  Arms: CAP Herbal Mint
Drug: CAP Mountain Berry — Sunscreen lip balm.
  Arms: CAP Mountain Berry
Drug: SPF Standard Sunscreen — SPF Standard (7 percent [%] Padimate-O and 3% Oxybenzone)
  Arms: SPF Standard

SUMMARY:
The purpose of this study is to determine the 80-Minute Water Resistant SPF of three sunscreen products (ChapStick Active Performance [CAP] UnScented, CAP Herbal Mint Flavour and CAP Mountain Berry Flavour) using the methodology described in the Food and Drug Administration (FDA) Final Rule (2011).

DETAILED DESCRIPTION:
A single-center, randomized, controlled, intra-individual comparison, evaluator-blind, clinical study to determine the 80-minute water resistant SPF of three sunscreen lip balms. Each participant will evaluate two of the three test products, an SPF standard and no treatment. Study treatments will be randomly assigned to 4 test sites delineated on the skin of the participant's back. The two test products will be applied to their allocated test sites prior to the 80-minute water immersion procedure (four 20-minute water immersion periods, each followed by a 15-minute air-drying period); the SPF standard will be applied to its allocated test site on completion of the final air-drying period. Test sites will be exposed to doses of ultraviolet (UV) radiation and erythemal response evaluated 16-24 hours later. Minimal erythema dose (MED) will be determined for protected and unprotected sites and used to determine the SPF value of each test product.

ELIGIBILITY:
Inclusion Criteria:

* Participant must provide a signed and dated, legally effective, informed consent document, which indicates they have been informed of all pertinent aspects of the study, before any study procedures are performed.
* Participant must provide relevant details of their medical history and current/recent medications and treatments (self-reported).
* Participant must have completed an annual Health Insurance Portability and Accountability Act (HIPAA) Authorization form.
* Participant must have completed a Photo Release Form.
* Participant must be able to read, write, speak and understand English.
* Participant must be in good general health.
* Participant must have uniform skin color over the test area (skin of the back between the shoulder blades and above the waistline) and an ITA value more than (>)28 degree.
* Participant must have Fitzpatrick Skin Type I, II or III.
* Participant must have sufficient area of suitable skin on their back for at least six 40 square centimeter (cm^2) test sites.
* Willing to have body hair clipped by a technician if participant has excessive hair in the test area.
* Willing and able to complete the 80-minute immersion procedure (that is, four 20-minute immersions followed by four 15-minute air drying periods).
* Participant must have a valid form of personal identification (photo identity [ID], driver's license, passport, permanent resident card, military ID card; forms cannot be expired).
* Male and female participants of child-bearing potential must agree to use a highly effective method of contraception for the duration of the study and for 14 days after their last treatment application. (Note: A participant is considered to be of child-bearing potential if, in the opinion of the Principal Investigator [PI], they are biologically capable of having children and sexually active).

Exclusion Criteria:

* Participant with a scheduled or planned Covid-19 vaccination during likely dates of study participation.
* Participant with a history of abnormal response to sunlight/UV radiation.
* Participant with a history of sensitivity to any ingredient of the test material or skin marker pen, or to latex; or any known sensitivities/allergies, including but not limited to cosmetic/toiletry products and topically applied skin treatment products/drugs.
* Participant with any significant dermatological condition, such as atopic dermatitis (eczema), psoriasis, skin cancer, melanoma, active dermal lesions, nevi, blemishes or moles, lupus, diabetes, or connective tissue disease, that would increase the risk associated with participation. (Note: presence of non-dysplastic nevi, blemishes, or moles would be acceptable if, in the opinion of the PI, they will neither jeopardize participant safety or compromise study outcomes. A participant with dysplastic nevi should be disqualified).
* Participant receiving any treatment with medications that would, in the opinion of the PI, confound study outcomes or increase the risk associated with participation, such as systemic or topical corticosteroids, antibiotics, anti-inflammatory drugs, antihistamines, antihypertension medications, or any other photosensitive medications. (Note: The prohibited medication list will be available to site staff for reference during screening).
* Participant who has used topical or systemic steroids, antihistamines, antibiotics or anti-inflammatory medications within 7 days of Study Day 1 which, in the opinion of the PI, could interfere with study outcomes.
* Participant who has used/applied any personal care products (for example, lotions, sunscreens, sunless tanners) and/or topical medications in/on the test area within 24 hours of Study Day 1.
* Participant who is unwilling to cease use of personal care products (for example, lotions, sunscreens, sunless tanners) and/or topical medications in/on the test area for the duration of the study.
* Participant with any known communicable disease(s) (e.g. Human Immunodeficiency Virus [HIV], Sexually Transmitted Diseases [STD's], Hepatitis B, Hepatitis C, and so on).
* Participant with skeletal protrusions and/or extreme areas of curvature in the test area.
* Participant with a medical treatment/vaccination (other than the Covid-19 vaccination) planned during the study, which would make them ineligible, place them at undue risk, or confound the outcome of the study, per the discretion of the PI.
* Participant who has undergone any surgical procedure in the last 12 months.
* Participant who has undergone chemical or physical treatment procedures in the test area within the last 12 months.
* Planned hospitalization during the study.
* Participant who exceeds a weight limit of 300 pounds due to equipment limitations.
* Participant with any condition that might confound the study results, increase the risk associated with participation, or interfere with study participation.
* Female participant who is pregnant, planning to become pregnant during the study, or breastfeeding (self-reported).
* Participant with any visible sunburn or suntan in test area.
* Participant with visible sun damage, scarring or tattoos in the test area that would interfere with study participation.
* Participant with any sun exposure and/or use of an artificial tanning lamp on the test area within 2 months of Study Day 1.
* Participant who is unwilling to avoid sun exposure and/or cease use of an artificial tanning lamp on the test area for the duration of the study.
* Participant who has participated in any clinical study involving UV exposure within the last 2 months, or any other type of clinical study within the last 1 month.
* Participant who is an employee/contractor or immediate family member of the PI, study site or Sponsor.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2021-12-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoint and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at single center in United States.
Units Other Than Participants: back test sites
Groups:
- All Study Participants: Study participants were randomly assigned to receive a single topical application of up to 4 study treatments (CAP UnScented; CAP Herbal Mint; CAP Mountain Berry and SPF Standard) + 1 untreated site; 80+/-2 milligrams (mg) product was applied to each 40 square centimeter(cm^2) test site (2.00+/-0.05 mg/cm^2). 15-minutes (mins) after test product application, the participant was seated in a water tub, with their upper back submerged for four 20-mins immersions, each of which was followed by a 15-mins air drying period. After completing the final air-drying period, 80+/-2 mg (2.0 mg/cm^2+/-0.05 mg/cm^2) of the SPF standard (7 percent [%] Padimate-O and 3% Oxybenzone) was applied to its designated test site. Test sites received a progressive sequence of timed ultraviolet (UV) radiation exposures and were evaluated for erythema immediately after irradiation and 16-24 hours later. When one site was invalid the data set was removed from the SPF testing.
Period: Overall Study
Arm/Group | All Study Participants
Started | 15; 60 back test sites
CAP UnScented | 10; 10 back test sites (10 participants received CAP UnScented (10 test sites) of which 8 participants completed the study and 6 had test sites which were deemed to be invalid.)
CAP Herbal Mint | 12; 12 back test sites (12 participants received CAP Herbal Mint (12 test sites) of which 10 participants completed the study and 5 had test sites which were deemed to be invalid.)
CAP Mountain Berry | 8; 8 back test sites (8 participants received CAP Mountain Berry (8 test sites) of which 6 participants completed the study and of these 6 had test sites which were deemed to be invalid.)
SPF Standard | 15; 15 back test sites
Untreated Sites | 15; 15 back test sites
Completed | 12; 32 back test sites
Not Completed | 3; 28 back test sites
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: Safety Population: all randomized participants who received at least one dose of a study treatment.
Groups:
- All Study Participants: Study participants were randomly assigned to receive a single topical application of up to 4 study treatments (CAP UnScented; CAP Herbal Mint; CAP Mountain Berry and SPF Standard) + 1 untreated site; 80+/-2 mg product was applied to each 40 cm^2 test site (2.00+/-0.05 mg/cm^2). 15-mins after test product application, the participant was seated in a water tub, with their upper back submerged for four 20-mins immersions, each of which was followed by a 15-mins air drying period. After completing the final air-drying period, 80+/-2 mg (2.0 mg/cm^2+/-0.05 mg/cm^2) of the SPF standard (7% Padimate-O and 3% Oxybenzone) was applied to its designated test site. Test sites received a progressive sequence of timed UV radiation exposures and were evaluated for erythema immediately after irradiation and 16-24 hours later. When one site was invalid the data set was removed from the SPF testing.
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0
  18 to 70 years | 12
  >70 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
  Unknown | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Arithmetic Mean SPF Values
Description: SPF values for each test product and the SPF standard were first calculated for each individual participant:SPFi = MEDp/MEDuR (p=protected [treated] site; u=unprotected [untreated] site). The arithmetic mean SPF, standard deviation (SD) and standard error (SE) were then calculated separately for each test product and the SPF standard from valid SPFi data: SPF = (ΣSPFi)/n; SD = √[(ΣSPFi^2) - ((ΣSPFi)^2/n) /(n-1))]; SE = SD/√n (n = no. participants providing valid test results). For SPF determination to be considered valid, in compliance with FDA Final Rule 2011, the mean SPF value of the SPF standard should fall within the SD range of the expected SPF (i.e.,16.3 ± 3.43 or 12.87 to 19.73).
Time Frame: From 16 to 24 hours post UV exposure
Population: Data could not be collected for primary outcome: required number of valid datasets (>=10) not achieved to calculate mean SPF
Groups:
- CAP UnScented: Participants with valid data for CAP UnScented.
- SPF Standard (CAP UnScented Dataset): Participants with valid data for SPF Standard (CAP UnScented dataset).
- CAP Herbal Mint: Participants with valid data for CAP Herbal Mint.
- SPF Standard (CAP Herbal Mint Dataset): Participants with valid data for SPF Standard (CAP Herbal Mint dataset).
- CAP Mountain Berry: Participants with valid data for CAP Mountain Berry.
- SPF Standard (CAP Mountain Berry Dataset): Participants with valid data for SPF Standard (CAP Mountain Berry dataset).
Arm/Group | CAP UnScented | SPF Standard (CAP UnScented Dataset) | CAP Herbal Mint | SPF Standard (CAP Herbal Mint Dataset) | CAP Mountain Berry | SPF Standard (CAP Mountain Berry Dataset)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From screening until 14 days after last dose administration of trial product (Up to 16 days)
Description: Adverse events (AEs), and therefore all serious adverse events (SAEs), were to be collected from immediately after a participant provided written consent to participate in the trial until 14 days after the last administration of study treatment (or the last study procedure). All SAEs were to be reported within 24 hours of detection. AEs were to be classified by Intensity (mild, moderate, severe); Causality (probable, possible, unlikely); Seriousness (serious or non-serious).
Arm/Group | CAP UnScented | SPF Standard (CAP UnScented Dataset) | CAP Herbal Mint | SPF Standard (CAP Herbal Mint Dataset) | CAP Mountain Berry | SPF Standard (CAP Mountain Berry Dataset)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/10 | 0/10 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/10 | 0/10 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/10 | 0/10 | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/99/NCT05124899/Prot_SAP_000.pdf